CLINICAL TRIAL: NCT03711396
Title: ENgaging in Advance Care Planning Talks Group Visit Intervention (ENACT) for Individuals With Amnestic Mild Cognitive Impairment (aMCI)
Brief Title: ENgaging in Advance Care Planning Talks Group Visit Intervention for Cognitive Impairment
Acronym: ENACT-aMCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-1459
Record Dates: First submitted 2018-10-11; First posted 2018-10-18 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Advance Care Planning
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: We will conduct four n-of-1 group visit interventions for advance care planning.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advance Care Planning Group Visits - amnestic Mild Cognitive Impairment (Experimental): Participants with amnestic Mild Cognitive Impairment will attend group visits to discuss advance care planning with their study partners. Group visits will last up to two hours and be help up to twice.
  Interventions: Behavioral: Advance Care Planning Group Visits
- Advance Care Planning Group Visits - Care Partners (Experimental): Care partners of persons with amnestic Mild Cognitive Impairment will attend group visits, with the person with Mild Cognitive Impairment, to discuss advance care planning. Group visits will last up to two hours and be help up to twice.
  Interventions: Behavioral: Advance Care Planning Group Visits

INTERVENTIONS:
Behavioral: Advance Care Planning Group Visits — Pilot test the Advance Care Planning Group Visit intervention adaptations, called ENgaging in Advance Care planning Talks Group Visit intervention (ENACT Memory Group Visits), to see if it is feasible, acceptable and improves the number of people with amnestic mild cognitive impairment who complete an advance directive (a legal form that describes someone's wishes for future medical care if they are unable to make their own decisions). It will also see how ready individuals are to participate in advance care planning. The overall goal is to improve opportunities for older adults with amnestic mild cognitive impairment to receive medical care that is consistent with their values, goals, and preferences.

SUMMARY:
The Advance Care Planning Group Visit intervention is a new intervention that uses the strengths of group visits to promote advance care planning conversations and documentation. However, the Advance Care Planning Group Visit intervention was initially designed for individuals without cognitive impairment. This study will specifically investigate ways to adapt the Advance Care Planning Group Visit intervention for individuals with amnestic Mild Cognitive Impairment and their family care partners.

DETAILED DESCRIPTION:
Advance care planning is a process that supports adults at any age or stage of health in understanding and sharing their personal values, life goals, and preferences regarding future medical care. The goal of advance care planning is to help ensure that people receive medical care that is consistent with their values, goals and preferences during serious and chronic illness.

The Advance Care Planning Group Visit intervention is a new intervention that uses the strengths of group visits to promote advance care planning conversations and documentation. However, the Advance Care Planning Group Visit intervention was initially designed for individuals without cognitive impairment. This study will specifically investigate ways to adapt the Advance Care Planning Group Visit intervention for individuals with amnestic Mild Cognitive Impairment.

This is a pilot test of the Advance Care Planning Group Visit intervention adaptations, called ENgaging in Advance Care planning Talks Group Visit intervention (ENACT Memory Group Visits), to see if it is feasible, acceptable and improves the number of people with amnestic mild cognitive impairment who complete an advance directive (a legal form that describes someone's wishes for future medical care if they are unable to make their own decisions). It will also see how ready individuals are to participate in advance care planning. The overall goal is to improve opportunities for older adults with amnestic mild cognitive impairment to receive medical care that is consistent with their values, goals, and preferences.

This aim will use rapid-cycle prototyping (n-of-1 interventions) to conduct the ENgaging in Advance Care planning Talks (ENACT) Memory Group Visits, adapting them for individuals with amnestic Mild Cognitive Impairment. Each n-of-1 prototype will include up to 10 patient-study partner dyads meeting in up to two 2-hour group medical visit sessions, one month apart. Four cohorts will be conducted so that approximately 40 participants are involved in the n-of-1 prototypes of the ENACT Memory Group Visit intervention. The intervention will be conducted based on an intervention manual that will be refined and adapted with input from patients, study partners, and the research team of multidisciplinary clinicians. Participants will receive the Colorado Medical Durable Power of Attorney form and other appropriate advance care planning resources for individuals with aMCI.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of amnestic mild cognitive impairment
* ability to provide consent
* have a study partner who has regular interaction with the patient

Exclusion Criteria:

* known prior diagnosis of deafness/hearing loss that would limit group discussion participation
* inability to travel to study location
* not having access to a phone for follow up
* not having an individual who is able to serve as a study partner to the patient
* normal cognitive screen based on SPMSQ

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCHealth, Aurora, Colorado
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lum HD, Jones J, Matlock DD, Glasgow RE, Lobo I, Levy CR, Schwartz RS, Sudore RL, Kutner JS. Advance Care Planning Meets Group Medical Visits: The Feasibility of Promoting Conversations. Ann Fam Med. 2016 Mar;14(2):125-32. doi: 10.1370/afm.1906. PMID 26951587
- [Background] Lum HD, Sudore RL, Matlock DD, Juarez-Colunga E, Jones J, Nowels M, Schwartz RS, Kutner JS, Levy CR. A Group Visit Initiative Improves Advance Care Planning Documentation among Older Adults in Primary Care. J Am Board Fam Med. 2017 Jul-Aug;30(4):480-490. doi: 10.3122/jabfm.2017.04.170036. PMID 28720629
- [Background] Lum HD, Dukes J, Daddato AE, Juarez-Colunga E, Shanbhag P, Kutner JS, Levy CR, Sudore RL. Effectiveness of Advance Care Planning Group Visits Among Older Adults in Primary Care. J Am Geriatr Soc. 2020 Oct;68(10):2382-2389. doi: 10.1111/jgs.16694. Epub 2020 Jul 29. PMID 32726475

RESULTS

PARTICIPANT FLOW:
Groups:
- Advance Care Planning Group Visits - aMCI: Participants with amnestic mild cognitive impairment (aMCI) will attend group visits to discuss advance care planning with their study partners. Group visits will last up to two hours and be held up to twice.
- Advance Care Planning Group Visits - Care Partners: Participants who are the care partners of persons with amnestic mild cognitive impairment (aMCI) will attend group visits (with the person with aMCI) to discuss advance care planning with their study partners. Group visits will last up to two hours and be held up to twice.
Period: Overall Study
Arm/Group | Advance Care Planning Group Visits - aMCI | Advance Care Planning Group Visits - Care Partners
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants with aMCI who were enrolled to group visits with a study partner. Demographics data were not collected for the care partners.
Groups:
- Intervention: Participants attended two group visits one month apart to discuss advance care planning and to receive information about advance care planning.
Arm/Group | Intervention
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.7 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
Education [Count of Participants; unit: Participants] — Highest level of education received by participant with aMCI
  Participants
    High School Graduate | 3
    Some College | 1
    College Graduate | 2
    Any Post-graduate | 7
Relationship status [Count of Participants; unit: Participants] — Current relationship status of participants with aMCI
  Participants
    Married/with partner | 10
    Widowed | 1
    Divorced/separated | 2
Caregiver in the last 12 months [Count of Participants; unit: Participants] — Has the participant with aMCI been the caregiver for another person in the last 12 months
  Participants
    Yes | 2
    No | 11
Self-Rated Health [Count of Participants; unit: Participants]
  Excellent | 8
  Good | 3
  Fair | 2
  Poor | 0
  Very Poor | 0
Relationship of Study Partner to Participant [Count of Participants; unit: Participants]
  Spouse | 9
  Partner | 1
  Child | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Readiness to Engage in ACP (ACP Engagement Scale)
Description: The Advance Care Planning (ACP) Engagement Scale will be used to assess readiness to engage in specific parts of the advance care planning process (i.e. signing official papers to name a medical decision maker; talking to the decision maker; talking to the doctor; signing official papers putting their wishes in writing). Items are rated on a Likert scale, with possible scores ranging from 1-5. Higher scores indicate a higher level of engagement with the advance care planning behavior and a better outcome.
Time Frame: 0, 3 months
Population: Participants with aMCI
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Advance Care Planning Group Visits - Persons With aMCI: Participants with amnestic Mild Cognitive Impairment will attend group visits to discuss advance care planning with their study partners. Group visits will last up to two hours and be help up to twice.
Arm/Group | Advance Care Planning Group Visits - Persons With aMCI
Number analyzed (Participants) | 13
units on a scale
  Readiness to sign official papers naming a medical decision maker at 0 months | 1.92 (1.12)
  Readiness to talk to decision maker at 0 months | 1.54 (0.88)
  Readiness to talk to doctor at 0 months | 2.77 (1.36)
  Readiness to sign papers putting wishes into writing at 0 months | 2.00 (1.15)
  Readiness to sign official papers naming a medical decision maker at 3 months | 1.77 (0.93)
  Readiness to talk to decision maker at 3 months | 2.38 (0.96)
  Readiness to talk to doctor at 3 months | 2.00 (0.91)
  Readiness to sign papers putting wishes into writing at 3 months | 2.08 (1.16)

2. Secondary Outcome: Change in Readiness to Engage in ACP (ACP Engagement Score) - Care Partner Reported
Description: Care partner report of the Advance Care Planning (ACP) Engagement Scale will be used to assess care partner perspectives on the person with amnestic mild cognitive impairment's readiness to engage in specific parts of the advance care planning process (i.e. signing official papers to name a medical decision maker; talking to the decision maker; talking to the doctor; signing official papers putting their wishes in writing). Items are rated on a Likert scale, with possible scores ranging from 1-5. Higher scores indicate a higher level of engagement with the advance care planning behavior and a better outcome.
Time Frame: 0, 3 months
Population: Care partners of persons with aMCI
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Advance Care Planning Group Visits - Care Partners: Care partners of persons with amnestic mild cognitive impairment who participated in the advance care planning group visits.
Arm/Group | Advance Care Planning Group Visits - Care Partners
Number analyzed (Participants) | 13
units on a scale
  Readiness to sign official papers naming a medical decision maker at 0 months | 1.92 (1.19)
  Readiness to talk to decision maker at 0 months | 2.31 (1.25)
  Readiness to talk to doctor at 0 months | 2.62 (0.96)
  Readiness to sign papers putting wishes into writing at 0 months | 1.62 (0.77)
  Readiness to sign official papers naming a medical decision maker at 3 months | 1.69 (1.11)
  Readiness to talk to decision maker at 3 months | 2.54 (0.88)
  Readiness to talk to doctor at 3 months | 1.77 (.93)
  Readiness to sign papers putting wishes into writing at 3 months | 1.92 (0.95)

3. Other Pre Specified Outcome: Advance Care Planning Intervention Evaluation
Description: Investigator-developed 7-item evaluation to assess participant rating of intervention comfort in the group setting, usefulness, preference compared to one-on-one visits, and helpfulness of talking with others. Each item is rated from "strong disagree" to "strongly agree" on a 5-point Likert scale. Scores can range from 1-5 with a score of 5 being a better outcome. This scale has not been specifically named. It has been published in the included reference.
Time Frame: Following Session Participation, 15 minutes after completed
Population: Combined persons with aMCI and care partners groups
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Advance Care Planning Group Visits - Amnestic Mild Cognitive Impairment: Participants with aMCI completed an evaluation of the intervention prototype.
Arm/Group | Advance Care Planning Group Visits - Amnestic Mild Cognitive Impairment | Advance Care Planning Group Visits - Care Partners
Number analyzed (Participants) | 13 | 13
score on a scale
  Group setting is better for ACP discussion than normal doctor visit | 4.23 (1.09) | 4.69 (0.48)
  The group discussion gave me useful information | 4.62 (0.51) | 5.00 (0.00)
  I felt comfortable talking about ACP in the group setting | 4.54 (0.66) | 4.92 (0.28)
  Talking with other people about ACP was helpful | 4.23 (1.36) | 5.00 (0.00)
  I feel the group visit addressed my specific questions | 4.31 (0.75) | 4.46 (0.66)
  I feel able to discuss ACP with my regular healthcare provider | 4.62 (0.51) | 4.38 (0.65)
  I would recommend these group visit sessions to a friend | 4.38 (1.45) | 4.92 (0.28)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Advance Care Planning Group Visits: Participants will attend group visits to discuss advance care planning with their study partners. Group visits will last up to two hours and be help up to twice.
  Advance Care Planning Group Visit: Aim 1: The first part of this study will focus on refining and adapting the Advance Care Planning Group Visit intervention so that it meets the needs of persons with amnestic cognitive impairment and a study partner who participates with them.
  Aim 2: The second part of the study will pilot test the Advance Care Planning Group Visit intervention adaptations, called ENgaging in Advance Care planning Talks Group Visit intervention (ENACT Memory Group Visits), to see if it is feasible, acceptable and improves the number of people with amnestic mild cognitive impairment who complete an advance directive (a legal form that describes someone's wishes for future medical care if they are unable to make their own decisions). It will also see how ready individuals are to participate in advance care planning. The overall goal is to improve opportunities for older adults with amnestic mild cognitive impairment to receive medical care that is consistent with their values, goals, and preferences.
Arm/Group | Advance Care Planning Group Visits
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT03711396/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT03711396/SAP_001.pdf
  • Informed Consent Form (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT03711396/ICF_002.pdf